CLINICAL TRIAL: NCT02267096
Title: Lombardi Comprehensive Cancer Center/Legacy Pilot Study to Reduce Adverse Smoking Outcomes in the Context of Lung Cancer Screening
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Prevent Cancer Foundation (Other)
Responsible Party: Principal Investigator, Kathryn L. Taylor, Ph.D., Professor, Department of Oncology, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-541
Record Dates: First submitted 2014-10-07; First posted 2014-10-17 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Smoking; Lung Cancer
Keywords: lung cancer screening
MeSH Terms: conditions — Smoking; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telephone Counseling (TC) (Experimental): The TC arm will receive the list of minimal treatment interventions plus 3-6 sessions of stepped-care, proactive, telephone counseling.
  Interventions: Behavioral: Telephone Counseling; Behavioral: Minimal Treatment
- Minimal Treatment (Active Comparator): The minimal treatment intervention includes a list of print, online, national telephone quitline phone number, and in-person cessation resources that is sent to participants.
  Interventions: Behavioral: Minimal Treatment

INTERVENTIONS:
Behavioral: Telephone Counseling — The TC arm includes a stepped care approach, 3-6 phone sessions, depending on each participant's needs. Within 1-2 days post-T1 assessment, the intervention will begin. Sessions 1-3 (15 min each) will occur approximately weekly over 3-4 weeks, scheduled at participants' convenience and at strategic therapeutic times (e.g., shortly pre/post-quit date). Continuing smokers or newly quit former smokers who would benefit from relapse prevention sessions will receive up to 3 additional sessions, to be completed within 3-4 weeks. The provision of 3-6 sessions is more intensive than several other telephone counseling interventions. A dose response relationship between quitting and number of sessions has been shown in non-volunteer smokers, and based on our pilot data, the investigators expect that a more intensive intervention will be needed for some participants.
  Arms: Telephone Counseling (TC)
Behavioral: Minimal Treatment — A list of self-help materials (print-, web-, phone-based), the national telephone quitline phone number, and local in person cessation resources will be given to all participants.

SUMMARY:
In 2011, the National Lung Screening Trial (NLST) reported that lung cancer mortality was reduced by 20% with spiral computed tomography (CT) compared to chest X-ray. It is estimated that 8 million people in the US are at high risk for lung cancer and that lung screening could prevent 12,000 deaths annually. Cost effectiveness models suggest that concurrent smoking cessation programs will be essential in order to realize the full benefit of screening. However, there are no clinical guidelines or evidence-based cessation protocols with demonstrated effectiveness in this setting. The investigators are addressing this gap by rigorously testing whether two scalable and pragmatic interventions can significantly boost intention to quit and cessation rates.

DETAILED DESCRIPTION:
Although abstinence from tobacco remains the best method of lung cancer prevention, recent evidence from the National Lung Screening Trial indicated that lung cancer mortality was reduced by 20% with spiral computed tomography (CT) compared to chest X-ray. As a result, the United States Preventive Services Task Force now recommends lung cancer screening for high risk individuals (long-term current and former smokers, 55-80 years old). It is estimated that 8 million people in the US are at high risk and that lung screening could prevent 12,000 deaths annually. Cost effectiveness models suggest that concurrent smoking cessation programs will be essential in order to realize the full benefit of screening. However, there are no clinical guidelines or evidence-based cessation protocols with demonstrated effectiveness in this setting. The investigators propose to address this gap by rigorously testing whether two scalable and pragmatic interventions (minimal and moderate in intensity) can significantly boost intention to quit and cessation rates. The investigators will capitalize on the critical 'teachable moment' of learning of one's screening result. Incorporation of an individual's screening result into a cessation intervention will test the innovative question of whether intention to quit can be enhanced and reduced intention to quit can be minimized, when an individualized, motivational telephone-based intervention is provided. Method: The investigators will accrue current smokers from the lung cancer screening programs at three sites: Georgetown University Hospital, Lahey Hospital, and Hackensack University Hospital. Prior to screening, 100 participants will be consented, enrolled, and will complete the baseline (T0) phone interview. Within 1-2 days of receiving the result, participants will be randomly assigned to Minimal Treatment (MT) vs. Telephone Counseling (TC). Both arms will receive the minimal treatment intervention (a list of print, online, quitline, and in-person cessation resources). The TC arm will receive 3-6 sessions of stepped-care, proactive, telephone counseling with the same Tobacco Treatment Specialist for both sites. Both arms will be assessed at 3-months post randomization for tobacco use outcomes. The specific aims are: 1) To conduct a two-arm randomized cessation intervention trial (MT vs. TC) with current smokers undergoing screening. 2) The investigators will explore moderators and mediators of the interventions' effect on cessation outcomes. Moderators include the screening result, race, gender, age, and nicotine dependence. Mediators include teachable moment factors, baseline intention to quit, and process measures. Summary: This proof of concept study will determine intervention feasibility, effect sizes needed for a larger study, and potential moderators and mediators of the intervention. The long-term goal is to evaluate the intervention in a multisite trial and ultimately, to disseminate it for use by lung cancer screening programs. The innovation of this proposal is in joining disease prevention (smoking cessation) with early detection in a medical setting that has relevance for a substantial proportion of current smokers, suggesting that even a small increase in cessation has the potential for a very large public health benefit.

ELIGIBILITY:
Inclusion Criteria:

1. 55-80 years old
2. current smoker
3. > 30-pack years
4. English-speaking
5. ability to provide meaningful consent
6. enrolled to undergo lung cancer screening. -

Exclusion Criteria:

1. history of lung cancer
2. current treatment for other cancer -

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2014-01; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Smoking Status with biochemical verification | Measured at 3 months post-randomization
  Self-reported 7-day and 30-day point prevalence abstinence with biochemical verification among those who report having quit smoking.

SECONDARY OUTCOMES:
Timeframe of Participants' Intention to Quit Smoking | Measured at each assessment: baseline (T0), 1-2 days post-receipt of screening result (T1), one-month post-randomization (T2), and 3 months post randomization (T2)
  At each assessment, the investigators will ask for the timeframe of participants' intention to quit smoking. The question is worded as: "Next are statements that smokers and former smokers have said about quitting. Please tell me which statement best represents what you think right now."
  1____ I enjoy smoking so much I will never consider quitting no matter what happens 2 ____ I never think about quitting but I might someday 3 ____I rarely think about quitting and have no specific plans to quit 4 ____I sometimes think about quitting but have no specific plans to quit 5 ____I often think about quitting but have no specific plans to quit 6 ____I plan to quit in the next 6 months 7 ____I plan to quit in the next 30 days 8 ____I have already begun to cut down and I have set a quit date
Quit attempts | Measured at each assessment: baseline (T0), 1-2 days post-receipt of screening result (T1), one-month post-randomization (T2), and 3 months post randomization (T2)
  The questions are worded as follows:
  1. "How many times since our last interview have you quit smoking for 24 hours or longer?"
  2. "What was the LONGEST period of time that you were able to not smoke cigarettes at all since the last interview?"
Cigarettes per day | Measured at each assessment: baseline (T0), 1-2 days post-receipt of screening result (T1), one-month post-randomization (T2), and 3 months post randomization (T2)
  The question is worded as follows: "Since our last interview, on average, how many cigarettes per day did you smoke?"
  1. i did not smoke since the last interview
  2. less than one per day
  3. 1 per day
  4. 2-5 per day
  5. 6-10 per day
  6. 11-20 per day
  7. 20 per day
  8. 21-40 per day
  9. 41-60 per day
  10. more than 3 packs per day

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Hackensack University Medical Center, Hackensack, New Jersey

REFERENCES:
- [Background] Taylor KL, Cox LS, Zincke N, Mehta L, McGuire C, Gelmann E. Lung cancer screening as a teachable moment for smoking cessation. Lung Cancer. 2007 Apr;56(1):125-34. doi: 10.1016/j.lungcan.2006.11.015. Epub 2006 Dec 28. PMID 17196298
- [Background] Barry SA, Tammemagi MC, Penek S, Kassan EC, Dorfman CS, Riley TL, Commin J, Taylor KL. Predictors of adverse smoking outcomes in the Prostate, Lung, Colorectal and Ovarian Cancer Screening Trial. J Natl Cancer Inst. 2012 Nov 7;104(21):1647-59. doi: 10.1093/jnci/djs398. Epub 2012 Oct 26. PMID 23104210
- [Background] Tammemagi MC, Berg CD, Riley TL, Cunningham CR, Taylor KL. Impact of lung cancer screening results on smoking cessation. J Natl Cancer Inst. 2014 May 28;106(6):dju084. doi: 10.1093/jnci/dju084. Print 2014 Jun. PMID 24872540
- [Derived] Taylor KL, Hagerman CJ, Luta G, Bellini PG, Stanton C, Abrams DB, Kramer JA, Anderson E, Regis S, McKee A, McKee B, Niaura R, Harper H, Ramsaier M. Preliminary evaluation of a telephone-based smoking cessation intervention in the lung cancer screening setting: A randomized clinical trial. Lung Cancer. 2017 Jun;108:242-246. doi: 10.1016/j.lungcan.2017.01.020. Epub 2017 Feb 15. PMID 28216065